CLINICAL TRIAL: NCT04836052
Title: Omega-3 Oil Use in COVID-19 Patients in Qatar: a Randomized Controlled Trial
Brief Title: Omega-3 Oil Use in COVID-19 Patients in Qatar
Acronym: Omega3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRC-04-20-1120
Record Dates: First submitted 2021-03-14; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3-oil arm (Experimental): patients admitted to ICU in HMC on any kind of oxygen support will get omega-3-oil 2 gm PO/NGT/OGT twice daily for 28 days or till ICU discharge or till death .
  Interventions: Drug: Omega 3 fatty acid
- standard of care arm ( no omega -3-oil ) (No Intervention): patients admitted to ICU in HMC on any kind of oxygen support will get ( standard of care= No Omega-3-oil ) but their labs will be monitored

INTERVENTIONS:
Drug: Omega 3 fatty acid — omega-3-oil 2 gm twice daily PO/NGT/OGT for 28 days or ICU discharge or death.
  Arms: omega-3-oil arm

SUMMARY:
COVID-19 infection has been widely spread since December 2019 and causing many comorbidities and fatalities. The most common clinical presentation of COVID-19 patients admitted to ICUs is respiratory failure , hypoxia and acute lung injury.

While new therapies and vaccines are urgently being investigated, they may take an inordinate time to get to right people. Omega-3-oil has been shown to have less proinflammatory mediators that may have immunomodulating, anti-inflammatory and antiviral effect. Two main fatty acids in omega-3-oil including eicosapentaenoic acid and docosahexaenoic acid have shown benefit in patients with ARDS as well.

So, the investigators proposed a randomized controlled study to evaluate the effectiveness of omega-3-oil supplementation 2 gm PO/NGT/OGT twice daily for 28 days or till discharge or till death in COVID-19 critically ill patients admitted to ICU who require oxygen support.

DETAILED DESCRIPTION:
The outbreak of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) due to a novel coronavirus (COVID-19) has emerged from Wuhan, China in late December 2019 and spread rapidly worldwide. Until July 16, 2020, there has been more than 13 million confirmed cases worldwide and ~580,000 deaths attributed to the disease. With the fast evolution of this worldwide public-health emergency, the general public has demanded the urgent investigation of potentially beneficial drugs that may improve the outcome of those affected by SARS-CoV-2 infection. While new therapies and vaccines are urgently being investigated, they may take an inordinate time, or never be identified. In the world today, there is only one drug approved by the FDA for COVID-19 (Remdesivir), while the investigation of several other re-purposed drugs is potentially suggested for SARS-CoV-2 treatment. Many trials are taking place around the world, including some utilizing potentially dangerous drugs with considerable side effects and enormous costs. However, the clinical effectiveness and safety of all pharmacologic therapies so far have not been fully proven.

The preliminary findings about this disease indicates that patients with cardiovascular risk factors including diabetes, obesity and other pre-existing cardiovascular diseases have worse outcomes. Additionally, severe respiratory infection and hypoxia associate with severe COVID-19 might trigger many pathological pathways which leads to cardiovascular sequelae. In a cohort of 416 hospitalized patients with COVID-19, myocardial injury defined by an elevated high sensitivity troponin I level was associated with in-hospital mortality. Another study of 187 hospitalized patients with COVID-19 showed a similar association. Interestingly, the highest mortality rates were observed among patients with pre-existing cardiovascular disease. Importantly, none of the published experiences from anywhere in the world has explored omega-3 oil and its known protective cardiovascular benefits.

Omega-3 fatty acids are found in food such as fish and flaxseed as well as in dietary supplements labeled omega-3-oil.The beneficiary role of Omega-3 polyunsaturated fatty acids (PUFA), namely eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) from fish, other marine sources, and supplements, have been shown to be anti-inflammatory through several cellular mechanisms including their incorporation into cellular membranes and resulting altered synthesis of eicosanoids. There is the potential that arachidonic acid (AA,) eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), and other dietary unsaturated fatty acids can inactivate enveloped viruses. It is thought that these fatty acids and others cause leakages or lysis of the viral envelopes by disrupting the membrane integrity, amongst other potential mechanisms. Indeed, the supplementation of EPA and DHA raises the level of these fatty acids in the phospholipids of cells involved in inflammation in a time and dose-dependent fashion at the expense of AA4. Li and colleagues reviewed 89 systematic reviews and meta-analyses investigating fish intake and all-cause mortality, concluding that fish intake at 2-4 servings per week is associated with the largest risk reduction.

In animal models despite these potential positive effects, there is conflicting evidence in relation to fish or fish oil consumption for some viral infections. In influenza models, fish oil-fed mice demonstrated impaired resistance to influenza infection due to their immunomodulatory and anti-inflammatory properties, which negatively dampened the immune response of the mice against the infection. In another mouse model, fish oil intake delayed influenza virus clearance and impaired the immune response in the lungs of mice by disrupting interferon-γ and immunoglobulin A. A further study indicated that it may be due to the impairment of virus-specific T lymphocyte cytotoxicity.

Despite the potential benefit, there are few human studies with omega 3 and immune and inflammatory response. The recent proposed benefit for omeg-3-oil is unique, EPA and DHA which are main fatty acids in omega-3-oils may act as substrates for the synthesis of specialized pro-resolving lipid mediators such as maresins, resolvins, and protectins, of which protectins may reduce the replication of influenza and potentially affect the inflammatory manifestations of respiratory viral diseases.

Notably, an in vitro model of human cells (Huh-7 and VeroE6) infected with a human coronavirus (HCoV-229E) demonstrated that several bioactive lipids downstream of phospholipase A2 (PLA2) activation were upregulated by the host cells. It is postulated that coronaviruses modulate the host lipid profile to optimize and maintain a specific homeostasis for viral replication. However, exogenous supplementation of AA and linoleic acid suppressed viral replication by interfering with the optimal host lipid conditions for viral replication. Notably, exogenous supplementation of AA and linoleic acid was also conserved when human cells were infected with MERS. However, exogenous supplementation of AA and linoleic acid suppressed viral replication by interfering with the optimal host lipid conditions for viral replication. Notably, exogenous supplementation of AA and linoleic acid was also conserved when human cells were infected with MERS. EPA, DHA, and AA also inhibited the replication of enterovirus A71 and coxsackievirus A16.While it is suggested that the oral or intravenous administration of various bioactive lipids could potentially reduce the severity and/or enhance the recovery of those infected with COVID-19, a dietary prophylactic approach or a dietary strategy for recovering patients is also worth considering. Further research is certainly required, as increasing AA via the diet might seem counterintuitive, as it is mainly proinflammatory.

Other clinical research about several lung infections, found the administration of PUFA can improve the outcome of the patient in acute pneumonia. Recent study reported that the dietary supplementation of ω-3 PUFA can exert an overall beneficial effect against acute pneumonia through the upregulation of the host's specific and nonspecific immune defenses.

Inflammation resolution is strongly dependent on lipid mediators, the specialized pro-resolution mediators (SPMs). As mentioned above, omega-3 polyunsaturated fatty acids (n-3 PUFAs) are precursors of very potent SPMs, including resolvins, protectins and maresins. In addition, they are associated with a less aggressive inflammatory initiation, after competing with omega-6 fatty acids for eicosanoid synthesis. Therefore, it makes sense to consider the use of n-3 PUFAs for clinical management of COVID-19 patients.

Recent clinical studies In ARDS patients, the enteral use of n-3 PUFAs has been associated to oxygenation improvement, reduced duration of mechanic ventilation as well as shorter ICU length of stay. In another study, critically ill patients receiving parenteral nutrition therapy enriched with fish oil lipid emulsion (rich in n-3 PUFAs EPA and DHA) were reported to have decreased infection and sepsis risk (40% to 56%, respectively) and a reduction of length of hospital and ICU stay by about two day.

As eluded previously, 2 cohort studies from China indicate that a significant proportion of hospitalized patients with COVID-19 developed some degree of myocardial injury. Coronary atherosclerotic plaques are more prone to rupture in response to an exacerbated inflammatory response during SARS-CoV-2. The use of n-3 FA (4-6 g/d) for improving atherosclerotic cardiovascular disease risk in patients with hypertriglyceridemia is supported by a 25% reduction in major adverse cardiovascular events in REDUCE-IT.

Furthermore, several drugs will increase triglyceride concentrations in patients with underlying high triglycerides. The effects of n-3 FA on drug-induced HTG have received relatively little attention, but n-3 FAs have uniformly been reported to lower triglycerides when used with interferon-α, antipsychotics, l-asparaginase, oral estrogens, protease inhibitors, retinoic acid, and sirolimus. In contrast with COVID-19 there is scarce of information published till now about role of n-3 FAs.

Collectively, these findings suggest that omega-3 fatty acids have properties that could improve oxygenation and outcome of COVID-19 patients. The utilization of omega-3-oil as safe, available and inexpensive therapy could be a promising therapeutic approach against SARS-CoV-2. Moreover, recent analysis of 8 studies showed that consumption of omega 3 oil up to 10 gm per day is safe in ICU.

However, due to lack of sufficient clinical data supporting either the beneficial or harmful effects of omega-3 oil use in patients with COVID-19, the optimal strategy for the management of in COVID-19 is uncertain and remains to be elucidated - putting together all the known properties of omega 3 and what is known about the COVID-19, the investigators hypothesize that omega 3 could have a significant beneficial impact on the clinical outcome of infected patients. The aim of this study is to investigate in-hospital use of omega-3 oil and mechanical ventilator days, improvement in oxygenation, need for ventilator in non-ventilated patients, ICU- length of stay, hospital related length of stay, thrombosis, all-cause morbidity and mortality in COVID-19 patients in a in randomized prospective controlled trial.

There is no study or evidence on Omega 3 and COVID-19 infection and respiratory failure. The investigators propose a randomized controlled study to minimize the risk of bias and confounding factors.

ELIGIBILITY:
Inclusion Criteria:

1. adult ICU patients ≥18 years
2. confirmed COVID-19 infection
3. on-Oxygen support (mechanical ventilation, face masks, nasal cannula, etc.)
4. Previous history of omega-3-oil with discontinuation of at least 1 month prior to admission

Exclusion Criteria:

1. soya bean oil allergy
2. fish allergy
3. peanut allergy
4. fish oil allergy
5. pregnant women
6. Continuous use of Omega-3-oil till admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-08-24 (Estimated); Study Completion 2021-12-24 (Estimated)

PRIMARY OUTCOMES:
mechanical ventilator free days | 28 days
  28 minus (days patient spent on ventilator if successfully liberated from ventilator)

SECONDARY OUTCOMES:
Change in oxygenation | days 1, 3, 7
  PaO2/FiO2
Hospital Mortality | 28 days
  death during 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, DC, Qatar